CLINICAL TRIAL: NCT06244862
Title: JAK Inhibitor in Acquired Hemophagocytic synDrome in the Intensive Care Unit
Acronym: JAKAHDI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP220919
Record Dates: First submitted 2023-12-26; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2023-12

CONDITIONS: Hemophagocytic Syndromes
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Interventional medicinal product (Experimental)
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Oral ruxolitinib twice a day (10 mg x 2 during 28 days) in association with standard of care in HS.

SUMMARY:
Hemophagocytic syndrome (HS) is a rare condition that can be responsible for severe organ failure. Therapeutic guidelines are mainly based on observational studies and expert opinions: no therapeutic advance has been developed for years, explaining why mortality in HS remains high (Intensive Care Unit mortality ranging from 40 to 70%). If etoposide remains the gold standard in critically ill HS patients, nearly 20% of patients are refractory to this therapy: treatment escalation is common, most often requiring the administration of intensive treatments generating high toxicity. Ruxolitinib is the first approved JAK inhibitor. It has been associated with improvement of HS manifestations and survival in a pre-clinical murine model. Data in humans are scarce but promising.

The aim is to demonstrate that ruxolitinib, in association with standard of care, may reverse organ failure (as represented by Sequential Organ Failure Assessment (SOFA) score) better than standard of care alone in critically ill patients with acquired HS.

ELIGIBILITY:
Inclusion Criteria:

* adult patients older than 18 years
* acquired hemophagocytic syndrome, regardless of etiology, defined by the presence of 5 or 6 HLH-2004 criteria or HScore ≥ 200
* admission in the ICU
* need for symptomatic treatment of HS in relation with organ failure, as defined by SOFA score ≥ 4
* Informed consent signed:

  * by the patient,
  * Or informed consent signed by a family members/trustworthy person if his condition does not allow him to express his consent in written
* Or in an emergency situation and in the absence of family members/trustworthy person, the patient can be enrolled. The consent to participate to the research will be requested as soon as the condition of the patient will allow).
* The inclusion of women of childbearing potential requires the use of a highly effective contraceptive measure. Contraception should be maintained during treatment and one day after

Exclusion Criteria:

* Moribund, defined by a life expectancy < 48 hours;
* Pregnant or lactating patients (women of childbearing potential must have a negative urine or blood Human Chorionic Gonadotropin pregnancy test prior to trial entry);
* No affiliation to health insurance;
* Known hypersensitivity to ruxolitinib;
* Lactose intolerance;
* Hypersensitivity to cellulose, microcrystalline; magnesium stearate; silica, colloidal anhydrous; sodium starch glycolate (Type A); povidone K30; hydroxypropylcellulose 300 to 600 cps,
* Pre-existing decisions of withholding/withdrawing care,
* History of progressive multifocal leukoencephalopathy
* Uncontrolled cutaneous cancer
* Persons under psychiatric care that would impede understanding of informed consent and optimal treatment and follow-up
* Adults subject to a legal protection measure (guardianship, curatorship and safeguard of justice)
* Patients deprived of their liberty by a judicial or administrative decision
* Participation in another interventional research

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-08-08 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Survival with a decrease in SOFA score ≥ 3 points | At day 7
  Sequential Organ Failure Assessment Score varies from 0 to 4 and permit to assess organ failure. A higher score indicates better neurological function.

SECONDARY OUTCOMES:
Overall survival in HS critically ill patients | At 6 months
SOFA score | At day 1
  Sequential Organ Failure Assessment Score varies from 0 to 4 and permit to assess organ failure. A higher score indicates better neurological function.
SOFA score | At day 14
  Sequential Organ Failure Assessment Score varies from 0 to 4 and permit to assess organ failure. A higher score indicates better neurological function.
SOFA score | At day 28
  Sequential Organ Failure Assessment Score varies from 0 to 4 and permit to assess organ failure. A higher score indicates better neurological function.
Length of stay in Intensive Care Unit | Up to 6 months
  number of days in the ICU from inclusion to ICU discharge or death
Hospital length of stay | Up to 6 months
  number of days in the hospital from inclusion to hospital discharge or death
Measurement of clinical and biological manifestations | At day 1
  Measurements of temperature, ferritin level, CD25 soluble receptor dosage, fibrinogen level, triglycerides level, haemoglobin level, white blood cells count, platelets count
Measurement of clinical and biological manifestations | At day 7
  Measurements of temperature, ferritin level, CD25 soluble receptor dosage, fibrinogen level, triglycerides level, haemoglobin level, white blood cells count, platelets count
Measurement of temperature | At day 14
Measurement of temperature | At day 28
Measurement of ferritin level | At day 14
Measurement of ferritin level | At day 28
Measurement of CD25 soluble receptor dosage | At day 14
Measurement of CD25 soluble receptor dosage | At day 28
Measurement of fibrinogen level | At day 14
Measurement of fibrinogen level | At day 28
Measurement of triglycerides level | At day 14
Measurement of triglycerides level | At day 28
Measurement of haemoglobin level | At day 14
Measurement of haemoglobin level | At day 28
Measurement of white blood cells count | At day 14
Measurement of white blood cells count | At day 28
Platelets count | At day 14
Platelets count | At day 28
Dosages of IL2, IL6, IL10, IL12, GM-CSF, IFN gamma, TNF alpha | At day 1
Dosages of IL2, IL6, IL10, IL12, GM-CSF, IFN gamma, TNF alpha | At day 7
Dosages of IL2, IL6, IL10, IL12, GM-CSF, IFN gamma, TNF alpha | At day 14
Dosages of IL2, IL6, IL10, IL12, GM-CSF, IFN gamma, TNF alpha | At day 28
Incidence of nosocomial infections (viral and bacterial) | Until day 28
Incidence of adverse event, severe adverse event | Until day 28
  Intensity and frequency of adverse event and severe adverse event according to the CTCAE Toxicity Grading Scale for Determining The Severity of Adverse Events

IPD SHARING:
Plan to Share IPD: Undecided